CLINICAL TRIAL: NCT04969614
Title: Safety and Immunogenicity of 2-dose Inactivated COVID-19 Vaccine in Kidney Transplant Recipients: a Prospective Cohort Study
Brief Title: Safety and Immunogenicity of 2-dose Inactivated COVID-19 Vaccine in Kidney Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Tao Lin, West China Hospital, West China Hospital
Other Study IDs: WestChina-COVID
Record Dates: First submitted 2021-07-19; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Kidney Transplantation; SARS-CoV-2 Acute Respiratory Disease; Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- kidney transplant recipients: kidney transplant recipients receiving inactivated SARS-CoV-2 vaccine

SUMMARY:
The severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) has a major impact on transplant recipients, with mortality rates up to 20%. However, immunocompromised individuals have been excluded from studies of SARS-CoV-2 vaccines. In such patients, the immune response to vaccination may be blunted. To better understand the immunogenicity of SARS-CoV-2 vaccines in transplant recipients, we quantified the humoral response to SARS-CoV-2 vaccine in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

Receiving kidney transplantation in West China Hospital, Sichuan University

Exclusion Criteria:

1) History of rejection or infection over the previous 3 months; 2) receiving kidney transplantation >3 months; 3) Combined with HBV/HVC/HIV infection in the donor or recipient; 4) Malignancy history in the donor and recipient; 5) organ transplant history in the recipient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients receiving kidney transplantation in West China Hospital between 01/01/2015 and 01/03/2021
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
seropositive anti-COVID-19 antibody | 2 to 6 weeks after the second injection of inactivated vaccine
  seropositive anti-COVID-19 antibody, including IgM, IgG, and IgA